CLINICAL TRIAL: NCT04508413
Title: An Exploratory, 14-week, Open-label Clinical Food Study to Evaluate the Effects of KB295 in Adult Patients With Ulcerative Colitis (UC) Presenting With Mild-to-moderate UC Symptoms
Brief Title: A Clinical Study to Assess the Effects of KB295 in Patients With Ulcerative Colitis (UC) on Gut Microbiota Structure and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K030-120
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Ulcerative Colitis
Keywords: Microbiome; Ulcerative Colitis; Kaleido; Kaleido Biosciences; KB295; Oligosaccharide; Glycan; Pathogens; Microbiome metabolic therapy; MMT; Mild-to-moderate UC
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KB295 (Other)
  Interventions: Other: KB295

INTERVENTIONS:
Other: KB295 — KB295 is a novel glycan

SUMMARY:
This exploratory, open-label clinical study aims to explore the effects of KB295, a novel glycan, on adult patients with ulcerative colitis (UC) presenting with mild-to-moderate UC symptoms

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, ≥18 and ≤75 years of age
* Confirmed diagnosis of UC (>6 months) by endoscopy
* Mild-to-moderate UC with at least 4 weeks of UC symptomatology prior to screening
* Stable medication regimen for at least 2 weeks prior to screening, if on medication for UC

Exclusion Criteria:

* Possible or confirmed diagnosis of Crohn's disease or indeterminate disease
* History of isolated distal proctitis
* Use of any antidiarrheal medications within the last 1 week prior to screening
* Antibiotic treatment within the past 28 days prior to screening
* Any non-UC related immunosuppressive medications other than purine analogs. Systemic corticosteroids including prednisone > 10 mg per day are excluded.
* Major intra-abdominal surgery related to the bowel within 24 weeks prior to the screening period and/or planned invasive surgery/hospitalization during the study
* Major medical comorbidities, or other conditions in the opinion of the PI, that might impact the patient's safety or compliance, or the interpretation of the study results
* Treatment with any other investigational drugs within 28 days prior to the screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing any treatment-emergent adverse events (TEAEs) | Day -1 to Day 84
Number of patients experiencing discontinuations due to adverse events (AEs) | Day -1 to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wingertzahn, PhD, Study Director — Kaleido Biosciences
Locations (3):
- United States (2):
  - Atlantia Food Clinical Trials, Chicago, Illinois
  - Elligo Health Research, Inc., Austin, Texas
- Atlantia Food Clinical Trials, Cork, Ireland